CLINICAL TRIAL: NCT00906139
Title: Propofol and Fentanyl Versus Midazolam and Fentanyl for Sedation During Diagnostic or Therapeutic Gastrointestinal Endoscopy in Cirrhotic Patients
Brief Title: Propofol and Fentanyl Versus Midazolam and Fentanyl for Endoscopy Sedation in Cirrhotic Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Lucianna Pereira da Motta Pires Correia, Federal University of São Paulo
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCorreia
Record Dates: First submitted 2009-05-20; First posted 2009-05-21 (Estimated); Last update posted 2009-05-25 (Estimated); Status verified 2009-05

CONDITIONS: Cirrhosis
Keywords: Propofol; Midazolam; Cirrhosis; Gastrointestinal endoscopy; Complications; Sedation
MeSH Terms: conditions — Fibrosis | interventions — Propofol; Midazolam; Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propofol (Active Comparator): To receive propofol (0.5 mg/kg up to 400 mg) and fentanyl (0.05 mg);
  Interventions: Drug: Propofol; Drug: Fentanyl
- Midazolam (Active Comparator): To receive midazolam (0.1 mg/kg) and fentanyl (0.05 mg).
  Interventions: Drug: Midazolam; Drug: Fentanyl

INTERVENTIONS:
Drug: Propofol — Propofol dose: 0.5 mg/kg up to 400 mg
  Arms: Propofol
Drug: Midazolam — Midazolam dose: 0.1 mg/kg
  Arms: Midazolam
Drug: Fentanyl — Fentanyl dose: 0.05 mg

SUMMARY:
The purpose of this study is to compare propofol associated with fentanyl versus midazolam plus fentanyl for sedation during diagnosis or therapeutic upper gastrointestinal endoscopy (UGE) in cirrhotic patients.

DETAILED DESCRIPTION:
UGE is often performed in cirrhotic patients for the diagnosis and treatment of portal hypertension complications. Current data suggests that propofol sedation may have advantages over benzodiazepines. However, there are few reports comparing propofol versus midazolam in patients with liver cirrhosis. The study's objective is to compare propofol associated with fentanyl versus midazolam plus fentanyl for sedation during diagnosis or therapeutic UGE in cirrhotic patients. A prospective randomized study will include cirrhotic patients (Child A, B or C and ASA 2 or 3), referred for diagnostic or therapeutic UGE, randomized for group I: propofol (0,5 mg/kg up to 400 mg) and fentanyl (0,05 mg); or group II: midazolam (0,1 mg/kg) and fentanyl. Sedation was performed by an exclusively dedicated gastroenterologist. Efficacy (completion of procedures), complications (hypoxemia, hypotension, arrhythmias) and recovery time (elapsed from the end of the procedure and discharge) will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis, any etiology
* ASA II or III
* Child A, B or C
* Age between 18 years and 75 years
* Patients that agree in participate of study and signed the contentment term

Exclusion Criteria:

* Schistosomiasis
* Recuse
* Hepatocellular carcinoma
* Contraindications to drugs
* ASA IV or V
* Hepatic encephalopathy, neurologic diseases
* Opioids, narcotics, MAO inhibitors or benzodiazepines use
* Alcohol abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2008-03; Primary Completion 2009-02 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
To compare propofol and fentanyl versus midazolam and fentanyl regarding safety and efficiency | Three months

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil